CLINICAL TRIAL: NCT03330366
Title: An 8 Week, Randomized, Double-blind, Placebo-controlled Crossover Clinical Trial of Allium Hookeri Root Extract on Anti-diabetic Effects
Brief Title: Effects of Allium Hookeri on Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CTCF2_2015_AH
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allium hookeri extract (Experimental): take two capsules per day (486 mg/day) for 8 weeks
  Interventions: Dietary Supplement: Allium hookeri extract
- Placebo (Placebo Comparator): take two capsules per day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Allium hookeri extract — take two capsules per day (486 mg/day) for 8 weeks
  Other Names: AH
  Arms: Allium hookeri extract
Dietary Supplement: Placebo — take two capsules per day
  Arms: Placebo

SUMMARY:
The researchers investigated the anti-diabetic effects of Allium hookeri root extract for Korean prediabetic participants.

DETAILED DESCRIPTION:
Allium hookeri root is widely consumed as a vegetable and herbal medicine in Asia. Although the antidiabetic activities of Allium hookeri have been documented in animal studies, the improved effects of Allium hookeri on human are not clear. Therefore, in this study, the researchers investigated whether Allium hookeri root extract could be effective in reducing the risk of type 2 diabetes in individuals with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Fasting glucose 100~126 mg/dl

Exclusion Criteria:

* Significant variation in weight (more 10%) in the past 3 months
* Treatment by hypoglycemic and hypolipidemic drug therapy within the past three months
* Type 1 diabetes or HbA1c>9.0%
* Cardiovascular disease
* Hypoglycemic agent, obesity medicine, and lipid lowering agent within past 6 months or blood sugar, obesity, and lipid improvement functional foods within past 2 monts
* Pregnancy or breast feeding

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2016-07-08 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Changes of blood glucose during OGTT | 8 weeks
  Changes of fasting and postprandial glucose during OGTT were assessed before and after the intervention

SECONDARY OUTCOMES:
Changes of blood insulin | 8 week
  Changes of blood insulin were assessed before and after the intervention
Changes of C-peptide | 8 week
  Changes of C-peptide were assessed before and after the intervention
Changes of HbA1c | 8 week
  Changes of HbA1c were assessed before and after the intervention

REFERENCES:
- [Derived] Park SH, Bae UJ, Choi EK, Jung SJ, Lee SH, Yang JH, Kim YS, Jeong DY, Kim HJ, Park BH, Chae SW. A randomized, double-blind, placebo-controlled crossover clinical trial to evaluate the anti-diabetic effects of Allium hookeri extract in the subjects with prediabetes. BMC Complement Med Ther. 2020 Jul 6;20(1):211. doi: 10.1186/s12906-020-03005-3. PMID 32631388